CLINICAL TRIAL: NCT00834145
Title: Effect of Normatec Pump for Relief of Leg Edema in Patients With Right Heart Failure: Short- Intermediate- and Long-Term Outcomes
Brief Title: Effect of Normatec Pump for Relief of Leg Edema in Patients With Right Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: David Blondheim, M.D., Hillel Yaffe Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 32/2008
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2009-02

CONDITIONS: Right Heart Failure; Cor Pulmonale
Keywords: Edema; Right heart failure; Cor pulmonale; Pump; Leg compression
MeSH Terms: conditions — Heart Failure; Pulmonary Heart Disease; Edema

ARMS (2):
- 1 (Experimental): Patients will receive a NormaTec pump and perform active pumping twice daily during hospitalization and thereafter once daily in addition to routine medical therapy.
  Interventions: Device: A mechanical compression pump
- 2 (No Intervention): Routine medical treatment

INTERVENTIONS:
Device: A mechanical compression pump — Patients in the experimental arm will receive a NormaTec pump which will be used twice daily during hospitalization and once daily on an ambulatory basis. A cuff is placed over the leg and a pneumatic system automatically compresses the leg according to predefined parameters of pressure, time etc.
  Other Names: NormaTec Pump
  Arms: 1

SUMMARY:
Mobilization of fluid from the legs with the Normatec pump in patients with right heart failure, may empty the "reservoir" in the legs from excessive fluid, enabling fluid overload to collect there rather than in the liver or in other third spaces. Thus, we hypothesize that patients will lose weight, feel better, look better, be less prone to infections in their legs and to congestion of the liver.

DETAILED DESCRIPTION:
The protocol will be divided into 2 parts:

1. The initial pumping phase will be an in-hospital study, short term study. Patients will be randomly assigned to conventional/conservative treatment or to pump therapy. Within 24 hours of admission patients assigned to pump therapy will be recruited for the study and will begin therapy according to the protocol outlined in the table below. These patients will not be given diuretics unless required to because of shortness of breath with suspected left heart failure. Individualized programs regarding pumping frequency and pump parameters will be set for each patient and will be adjusted during the first few days and maintained throughout the study unless there is a reason to modify them.

   Data on both the conventional/conservative and the pump arms of the study will be collected at similar intervals. The duration of the in-hospital period will not be extended because of the study and is expected to be 3-7 days.
2. An intermediate-term study in which the patients from the phase 1 study will be ambulatory. During this phase of the study the effect of continuous maintenance and optimization will be monitored. Patients will come to the hospital for their pumping session at which time the protocol tests will be performed. Patients that were assigned to the conventional/conservative arm in phase 1 will be examined as per protocol at 1, 2 and 3 weeks after admission but BNP levels will be repeated only after the 3rd week.
3. At 3 and 6 months after admission, the "long term" phase of the study, a systematic investigation regarding repeat hospitalizations and their causes will be carried out by telephone interview and by a review of admission data from hospital records.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients
* Adults
* Right heart failure secondary to pulmonary hypertension (cor pulmonale)
* Pronounced leg edema

Exclusion Criteria:

* Patients in sepsis
* Hemodynamically unstable
* Renal failure (creatinine >2 mg%)
* Deep vein thrombosis
* Pregnancy
* Psychiatric/noncompliant patients
* Patients who will not sign the informed consent form

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Patient weight | 3 and 6 months

SECONDARY OUTCOMES:
Leg circumference, Pulmonary pressures, Cardiac function | 3 and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hille Yaffe Medical Ceter, Hadera, Israel